CLINICAL TRIAL: NCT07087496
Title: Effects Of Mobile Augmented Reality Learning On Insulin Administration Knowledge And Skills Of Patients With Type 2 Diabetes
Brief Title: Mobile Augmented Reality Learning On Insulin Administration Knowledge And Skills Of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Hale SEZER, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IZBU-HEM-HS-1; Izmir Bakırçay University (Other: Izmir Bakırçay University)
Record Dates: First submitted 2025-07-04; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabete Type 2; Augmented Reality; Patient Education; Patient Education Materials
Keywords: diabete type 2; Augmented Reality; Patient Education; Subcutaneous injection
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is a quasi-experimental study with a pre-test and post-test design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention Group 1 (Experimental): The Intervention Group 1 were given education on insulin administration with a brochure
  Interventions: Other: insulin administration training with brochure
- Intervention Group 2 (Experimental): Intervention Group 2 were given education with "Mobile Augmented Reality (MAR)
  Interventions: Other: Insulin application training with mobile augmented reality

INTERVENTIONS:
Other: Insulin application training with mobile augmented reality — Intervention Group 2 (MAR group): Before the training, the participants were briefly informed about how the application would be performed, and their written consent was obtained. Before the insulin administration training was started, the MAR program was shown to them on the tablet by the researcher and the process steps containing QR codes prepared for insulin administration were provided on a blue flat surface and information was given about the use of the application, and a pre-test was administered to determine their knowledge levels on insulin administration. Then, the education application program prepared for insulin administration was opened and the patients were allowed to use it. The training application was performed 20-25 times. Then the post-test was administered to the participants immediately after the training. At the post-test, they were administered the Knowledge Test and Scale for Satisfaction with Patient Education.
  Other Names: Interventation group 2
  Arms: Intervention Group 2
Other: insulin administration training with brochure — The Intervention Group 1 (Brochure group): Before the training, the participants were informed about the study, and their written consent was obtained.
  Before insulin administration training, a knowledge test was given as a pre-test to determine the participants' knowledge levels on insulin administrations. After the pre-test, a 15-20 minute practical training was given using the brochure prepared for insulin administrations. Immediately after the training, the knowledge test and Scale for Satisfaction with Patient Education were administered as a post-test. After the post-test, the participants were asked to self-administer insulin. The insulin administration skills of the patients were assessed by the researcher using the Insulin Administration Skill Assessment Checklist. After the assessment, the participants were informed about their deficiencies, or incorrect performances.
  Arms: The Intervention Group 1

SUMMARY:
The goal of this study to determine the effectiveness of insulin administration with augmented reality on increasing the knowledge and skills of patients newly diagnosed with type 2 diabetes on insulin administrations, determining patients' satisfaction with education and comparing the following two strategies: education with the Mobile Augmented Reality and education with the brochure.

* Is Mobile augmented reality application effective on the knowledge scores and insulin application skills of patients with type 2 diabetes on insulin applications?
* Does training with a mobile augmented reality application affect patients' satisfaction with patient education?
* Other patients with type 2 diabetes were given insulin administration training with a brochure prepared by the researcher. All patients who participated in the study were evaluated for insulin administration knowledge and skills after the training.

DETAILED DESCRIPTION:
The study was aimed at determining the effectiveness of insulin administration with augmented reality on increasing the knowledge and skills of patients newly diagnosed with type 2 diabetes on insulin administrations, determining patients' satisfaction with education and comparing the following two strategies: education with the Mobile Augmented Reality and education with the brochure.

Methods: The study was conducted between November 1, 2023 and December 31, 2024 with patients newly diagnosed with type 2 diabetes who volunteered to participate in the study and were hospitalized in the first and second wards of the Internal Medicine Department of a state hospital (n=100).

In this quasi-experimental study with the pre-test and post-test design, the participants were allocated into two groups. While the participants in The Intervention Group 1 were given education on insulin administration with a brochure in line with the literature, the participants in the Intervention Group 2 were given education with "Mobile Augmented Reality (MAR)".

The data were collected using the "Individual Information Form", "Knowledge Test", "Scale for Satisfaction with Patient Education", and "Insulin Administration Skill Assessment Checklist".

ELIGIBILITY:
Inclusion Criteria:

* Being newly diagnosed with Type 2 diabetes at Izmir Bakırçay University Çiğli Training and Research Hospital,
* Not having received diabetes training,
* Not knowing the insulin application,
* Not having used augmented reality before,
* Being 18 years of age or older,
* Being able to use a smartphone.

Exclusion Criteria:

* To be diagnosed with Type 2 diabetes at Izmir Bakırçay University Çiğli Training and Research Hospital,
* To have received diabetes education,
* To be familiar with insulin application, -To have used augmented reality before,-
* To be under the age of 18
* To be unable to use a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Insulin administration knowledge Test | from pre-training to immediate post-training
  The test prepared by the researcher consists of 10 questions aimed at measuring the insulin administration knowledge levels of patients with type 2 diabetes. The content validity rate (CVR) for each question and the content validity index including all the questions were determined as 0.96. In the 10-question knowledge test, the higher the number of correct answers, the higher the score. It is assumed that the higher the score, the higher the level of knowledge about the subject. The minimum score is 1 and the maximum score is 10.It was aimed to evaluate the insulin application knowledge of patients diagnosed with type 2 diabetes who received training with mobile augmented reality and brochure after the training compared to before the training. It was expected that the mean knowledge scores of patients with Type 2 diabetes who received insulin administration training with mobile augmented reality would be higher than those who received training with brochures.
Insulin administration skills checklist | from pre-training to immediate post-training
  The 24-item checklist was developed by the researcher through the literature review to assess the patient's insulin administration skills.The checklist took its final form after expert opinions were obtained from nurse specialists using the Davis technique (1992). In the checklist, each correct step was scored as 2 points, each semi-completed step was scored as 1 point, and each step not completed at all was scored as 0 zero points. It was aimed to evaluate the insulin administration skills of patients with type 2 diabetes who received training with mobile augmented reality and brochure. It was expected that the mean skill scores of Type 2 diabetic patients who received insulin application training with mobile augmented reality would be higher than those who received training with brochure.

SECONDARY OUTCOMES:
Scale for Satisfaction with Patient Education | to immediate post-training
  This one-dimensional scale developed by Çiftçi et al. (2022) includes 30 items whose responses are rated on a five-point Likert-type scale (Strongly Disagree, Somewhat Agree, etc.). The mean score for the overall scale is calculated by summing the scores of all the items. The highest and lowest possible scores that can be obtained from the overall scale are 150 and 30, respectively. The Cronbach's α coefficient of the scale was calculated as 0.98 in Çiftçi et al.'s study (2022), and 0.85 in the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkadir Gül, Master, Principal Investigator — Izmir Bakırçay University Internal Medicine Nursing; Hale Sezer, PhD, Study Director — Izmir Bakırçay University Faculty of Health Science
Locations (1):
- İzmir Bakırçay University Çiğli Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The changes in the scores of insulin administration knowledge and skills of patients with type 2 diabetes before and after training and the satisfaction levels of patients with insulin administration training given with two different strategies will be given as a data set.
Supporting Information: Analytic Code
Time Frame: Beginning 1 year after publication of results
Access Criteria: Data in excell format will be shared with researchers who want to conduct meta-analysis using the raw data of the study.

REFERENCES:
- [Background] Yuan PM, Talent JM, Gracy RW. A tentative elucidation of the sequence of human triosephosphate isomerase by homology peptide mapping. Biochim Biophys Acta. 1981 Dec 29;671(2):211-8. doi: 10.1016/0005-2795(81)90136-7. No abstract available. PMID 7326265
- [Background] Ernould C, Dorchy H, Francois B, Geussens H, Hens G, Loeb H. [Guide for young diabetics]. Rev Med Liege. 1972 Jun 1;27(11):371-4. No abstract available. French. PMID 5041361
- [Background] Ashby FG, Boynton G, Lee WW. Categorization response time with multidimensional stimuli. Percept Psychophys. 1994 Jan;55(1):11-27. doi: 10.3758/bf03206876. PMID 8036090
- [Background] Omura S, Nakagawa A, Hashimoto H, Oiwa R, Iwai Y, Hirano A, Shibukawa N, Kojima Y. Virantmycin, a potent antiviral antibiotic produced by a strain of Streptomyces. J Antibiot (Tokyo). 1980 Nov;33(11):1395-6. doi: 10.7164/antibiotics.33.1395. No abstract available. PMID 7251481
- [Background] Gonzalez Fuente T, Calderon Ruiz AM, Martin Casabona N. [Peripheral tuberculous adenitis]. Med Clin (Barc). 1984 Nov 10;83(15):648. No abstract available. Spanish. PMID 6521519
- [Background] Chak A. How far have we come with ultrasound miniprobes? Endoscopy. 1999 May;31(4):329-32. doi: 10.1055/s-1999-21. No abstract available. PMID 10376463
- [Background] Shaw JM. Suspected cyanide poisoning in two goats caused by ingestion of crab apple leaves and fruits. Vet Rec. 1986 Sep 6;119(10):242-3. doi: 10.1136/vr.119.10.242. No abstract available. PMID 3765303
- [Background] Ciftci B, Avsar G, Sarialioglu A. A psychometric assessment on patient education: Developing a satisfaction scale. Perspect Psychiatr Care. 2022 Oct;58(4):2237-2245. doi: 10.1111/ppc.13052. Epub 2022 Feb 16. PMID 35170766
- [Background] Kurt Y, Ozturk H. The effect of mobile augmented reality application developed for injections on the knowledge and skill levels of nursing students: An experimental controlled study. Nurse Educ Today. 2021 Aug;103:104955. doi: 10.1016/j.nedt.2021.104955. Epub 2021 May 13. PMID 34051543
- [Background] Foronda, C.L., Crenshaw, N., Briones, P.L., Snowden, K., Griffin, M.A., Mitzova- Vladinov, G., 2020. Teaching and learning the skill of intubation using Telehealth glasses. Clin. Simul. Nurs. 40, 31-35. https://doi.org/10.1016/j.ecns.2019.12.005.
- [Background] Byrne PJ, Senk PA. Google Glass in Nursing Education: Accessing Knowledge at the Point of Care. Comput Inform Nurs. 2017 Mar;35(3):117-120. doi: 10.1097/CIN.0000000000000339. No abstract available. PMID 28277435
- [Background] Salem S, Cooper J, Schneider J, Croft H, Munro I. Student Acceptance of Using Augmented Reality Applications for Learning in Pharmacy: A Pilot Study. Pharmacy (Basel). 2020 Jul 21;8(3):122. doi: 10.3390/pharmacy8030122. PMID 32708150
- [Background] Foronda CL, Alfes CM, Dev P, Kleinheksel AJ, Nelson DA Jr, O'Donnell JM, Samosky JT. Virtually Nursing: Emerging Technologies in Nursing Education. Nurse Educ. 2017 Jan/Feb;42(1):14-17. doi: 10.1097/NNE.0000000000000295. PMID 27454054
- [Background] Van Krevelen, D. W. F., Poelman, R. (2010). A survey of augmented reality technologies, applications and limitations. International journal of virtual reality, 9(2), 1-20
- [Background] An, J., Poly, L.-P., Holme, T.A., 2020. Usability testing and the development of an augmented reality application for laboratory learning. J. Chem. Educ. 97 (1), 97-105. https://doi.org/10.1021/acs.jchemed.9b00453
- [Background] Kececi A, Toprak S, Kilic S. How Effective Are Patient Education Materials in Educating Patients? Clin Nurs Res. 2019 Jun;28(5):567-582. doi: 10.1177/1054773817740521. Epub 2017 Nov 6. PMID 29103313
- [Background] Aldridge MD. Writing and designing readable patient education materials. Nephrol Nurs J. 2004 Jul-Aug;31(4):373-7. PMID 15453229
- [Background] ADA: American Diabetes Assocation, (2023). Classification And Diagnosis Of Diabetes: Standarts Of Medical Care İn Diabetes - 2023. Diabetes Care. 43(1), 1-212. https://doi.org/10.2337/Dc23-Sint
- [Background] Dikici, İ., Havlioğlu S. (2020). Tip 2 Diyabetli Hastaların, Hasta Yakınlarının ve Bakım Veren Hemşirelerin Eğitim Gereksinimlerinin Q Metodu ile İncelenmesi. Gevher Nesibe Journal Of Medical And Health Sciences, 5(7), 101-107.
- [Background] Özbek, Y., Özgül E. (2023). Diyabetli Bireylerde Covıd-19 Tedavi ve Bakım Yönetimi. Balkan Sağlık Bilimleri Dergisi, 2(1), 21-26.
- [Background] Küçük, S., Uludasdemir, D., Karşıgil, P., Güven İ. (2023). Tip 2 Diyabet Hastalarında Sağlıklı Yaşam Biçimi Davranışlarının Belirlenmesi ve Diyabet Öz Yeterliliği. Türkiye Diyabet ve Obezite Dergisi, 7(2), 112-121.
- [Background] 1. TEMD: Türkiye Endokrinoloji ve Metabolizma Derneği, (2022). Diabetes Mellitus ve Komplikasyonlarının Tanı, Tedavi ve İzlem Kılavuzu 2022. Güncellenmiş 15. Baskı. Ankara, 2022
- See also: IDF Diabetes Atlas 11th Edition — https://diabetesatlas.org/resources/idf-diabetes-atlas-2025/